CLINICAL TRIAL: NCT00758420
Title: A Randomized, Single Blind, Placebo Controlled, Multicenter Study to Evaluate Efficacy and Safety of Polidocanol Injectable Foam for the Treatment of Symptomatic, Visible Varicose Veins With Saphenofemoral Junction (SFJ) Incompetence.
Brief Title: Randomized, Single Blind, Placebo Controlled, to Evaluate Efficacy and Safety of Polidocanol Injectable Foam for Treatment of Symptomatic, Visible Varicose Veins With SFJ Incompetence
Acronym: Pilot
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: VAP.VV013
Record Dates: First submitted 2008-09-22; First posted 2008-09-25 (Estimated); Results first posted 2014-03-24 (Estimated); Last update posted 2021-04-21 (Actual); Status verified 2021-04

CONDITIONS: Varicose Veins
Keywords: Varicose Veins
MeSH Terms: conditions — Varicose Veins

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Varisolve (polidocanol endovenous mircofoam)
  Interventions: Drug: Varisolve (Polidocanol Endovenous Microfoam)
- 2 (Placebo Comparator): Agitated saline
  Interventions: Drug: Agitated Saline

INTERVENTIONS:
Drug: Varisolve (Polidocanol Endovenous Microfoam) — 1% polidocanol, up to 15 mL, one treatment session (initially up to 30 ml, reduced to up to 15 ml in Amendment #2)
  Arms: 1
Drug: Agitated Saline — 10 u/mL normal heparinized saline solution, up to 20 mL, one treatment session
  Arms: 2

SUMMARY:
The purpose of this study is to evaluate the effectiveness of polidocanol injectable foam in the relief of symptoms, improvement of appearance, and overall effectiveness and safety in the treatment of varicose veins compared to placebo.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the efficacy of polidocanol injectable foam vs placebo treatments in relief of symptoms using two disease specific questionnaires, establishment of a minimally important difference (MID) for the questionnaires, improvement in the appearance of visible varicosities by a patient and medical assessments aided by pre and post treatment photographs, and a central independent assessor evaluating pre and post treatment photographs. In addition, the study will evaluate the efficacy of polidocanol injectable foam vs the placebo treatment in the elimination of SFJ reflux or occlusion of the treated vein, and to determine whether the placebo procedure blinds the patient to treatment assignment.

ELIGIBILITY:
Inclusion Criteria:

* Males and Females 18-65 years old
* VEINES Sym Score less than 75 points
* Varicose Vein clinical classification CEAP 2, 3, 4, or 5
* Incompetence of SFJ associated with incompetence of the GSV or other major accessory vein
* Superficial venous disease manifested by both symptoms and visible varicosities
* Ability to comprehend and sign an informed consent document and completed study questionnaires in English

Exclusion Criteria:

* Incompetence of the SSV which substantially contributes to the filling of visible varicose veins
* Current or previous Deep Vein Thrombosis
* Leg obesity
* Peripheral arterial disease in the leg to be treated
* Reduced mobility
* Planned prolonged travel with limited mobility with in 4 weeks of treatment
* History of pulmonary embolism or stroke
* Major surgery, prolonged hospitalization or pregnancy within 3 months
* Current anticoagulation therapy (within 7 days of enrollment)
* Participation in a clinical study involving a investigational product within 3 months
* Major co-existing disease or clinically significant laboratory abnormalities
* Known allergic response to polidocanol or heparin or severe and/or multiple allergic reactions
* Women of childbearing potential not using effective contraception one month prior to enrollment and/or unwilling to continue while on study
* Pregnant or lactating women
* Current alcohol or drug abuse

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2008-10; Primary Completion 2009-07 (Actual); Study Completion 2009-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janet Rush, MD, Study Chair — BTG International Inc.
Locations (5):
- United States (5):
  - Scottsdale, Arizona
  - New York, New York
  - Charlotte, North Carolina
  - Winston-Salem, North Carolina
  - Bellevue, Washington

REFERENCES:
- [Derived] Gibson K, Kabnick L; Varithena(R) 013 Investigator Group. A multicenter, randomized, placebo-controlled study to evaluate the efficacy and safety of Varithena(R) (polidocanol endovenous microfoam 1%) for symptomatic, visible varicose veins with saphenofemoral junction incompetence. Phlebology. 2017 Apr;32(3):185-193. doi: 10.1177/0268355516635386. Epub 2016 Jul 9. PMID 27013511
- See also: Study Website — http://www.veinstudy.com

RESULTS

PARTICIPANT FLOW:
Groups:
- Active Treatment: polidocanol injectiable foam 1%, up to 15 mL, one treatment session
- Placebo: Agitated saline
  Agitated Saline: 10 u/mL normal heparinized saline solution, up to 20 mL, one treatment session
Period: Overall Study
Arm/Group | Active Treatment | Placebo
Started | 39 | 38
Completed | 39 | 38
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Treated patients with a week 8 study assessment.
Groups:
- Placebo: Agitated Saline: 10 u/mL normal heparinized saline solution, up to 20 mL, one treatment session
- Polidocanol Injectable Foam, 1.0%: Polidocanol injectable foam 1%, up to 15 mL, one treatment session
- Total: Total of all reporting groups
Arm/Group | Placebo | Polidocanol Injectable Foam, 1.0% | Total
Number analyzed (Participants) | 38 | 39 | 77
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.9 (10.71) | 45.3 (10.75) | 45.1 (10.66)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32 | 30 | 62
  Male | 6 | 9 | 15
Baseline VCSS [Mean (Standard Deviation); unit: units on a scale] — The Venous Clinical Severity Score (VCSS) was determined by a study staff member blinded to treatment assignment, (i.e., the 'blinded assessor'). The VCSS rates 9 clinical characteristics of chronic venous disease (pain, varicose veins, venous edema, skin pigmentation, inflammation, induration, and number, duration, and size of ulcers) using Grades 0 to 3 (absent to severe). An additional 0 to 3 points are added for differences in use of compression therapy (compression and elevation) to produce a 30-point maximum flat scale.
  units on a scale | 6.0 (1.95) | 6.6 (2.05) | 6.3 (2.01)
CEAP Clinical classification [Number; unit: participants] — Patients were eligible for study if they had a clinical classification of C2-C5 as follows: C2 Varicose veins C3 Edema C4 Skin changes without ulceration C5 Skin changes with healed ulceration.
  participants
    C3 - Edema | 34 | 35 | 69
    C4 - Skin Change Without Ulceration | 4 | 2 | 6
    C5 - Skin Change With Healed Ulceration | 0 | 2 | 2
VVSymQ Score [Mean (Standard Deviation); unit: units on a scale] — The VVSymQ is a subset of the VEINES-Sym and consists of the 5 symptoms most relevant to patients. The raw score, which can range from 5 to 30, was transformed to a summary VVSymQ score that ranges from 0 (worst possible symptom health) to 100 (best symptom health) using the following formula: VVSymQ: (Transformed Score) = [(Raw Score) - 5] * 4
  units on a scale | 57.5 (27.97) | 52.6 (29.37) | 55.0 (28.60)
VEINES-Sym Score [Mean (Standard Deviation); unit: units on a scale] — The VEINES-Sym summary score includes 10 items; 9 venous symptoms (heavy legs, aching legs, swelling, night cramps, heat or burning sensation, restless legs, throbbing, itching, tingling sensation), rated on a 6-point scale of frequency and leg pain rated on a 6-point scale of intensity (very severe, severe, moderate, mild, very mild, none). It can range from 0 to 100, with a '0' score indicating all symptoms were present all of the time in the past week and a '100' score indicating none of the symptoms were present at any time in the previous week.
  units on a scale | 61.9 (26.05) | 59.3 (26.11) | 60.6 (25.94)

OUTCOME MEASURES:

1. Primary Outcome: The Absolute Change From Baseline Score for the VVSymQ (Total Score) at 8 Weeks
Description: The VVSymQ is a subset of the VEINES-Sym and consists of the 5 symptoms most relevant to patients. The raw score, which can range from 5 to 30, was transformed to a summary VVSymQ score that ranges from 0 (worst possible symptom health) to 100 (best symptom health) using the following formula: VVSymQ: (Transformed Score) = [(Raw Score) - 5] * 4.
Time Frame: Baseline to 8 weeks
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Groups:
- Placebo: agitated saline
Arm/Group | Placebo | Polidocanol Injectable Foam, 1.0%
Number analyzed (Participants) | 38 | 39
units on a scale | 16.7 (3.18) | 30.7 (3.04)

ADVERSE EVENTS:
Arm/Group | Placebo | Polidocanol Injectable Foam, 1.0%
Serious Adverse Events (participants affected / at risk) | 1/38 | 1/39
Other Adverse Events (participants affected / at risk) | 19/38 | 36/39
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=38) | Polidocanol Injectable Foam, 1.0% (N=39)
Transient ischemic attack (Nervous system disorders) | 1 (1) | 0 (0)
Sick sinus syndrome (Cardiac disorders) | 0 (0) | 1 (1) — unrelated to study drug. resulted from pacemaker placement.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=38) | Polidocanol Injectable Foam, 1.0% (N=39)
chest discomfort (General disorders) | 0 (0) | 2 (2)
edema (General disorders) | 0 (0) | 2 (2)
nasopharyngitis (Infections and infestations) | 1 (1) | 2 (2)
contusion (Injury, poisoning and procedural complications) | 2 (2) | 10 (10)
incision site complication (Injury, poisoning and procedural complications) | 1 (1) | 3 (3)
incision site hematoma (Injury, poisoning and procedural complications) | 3 (3) | 4 (4)
arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
groin pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
limb discomfort (Musculoskeletal and connective tissue disorders) | 1 (1) | 10 (10)
musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 4 (4)
pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 6 (6)
headache (Nervous system disorders) | 0 (0) | 4 (4)
paresthesia (Nervous system disorders) | 0 (0) | 2 (2)
pruritis (Skin and subcutaneous tissue disorders) | 5 (5) | 3 (3)
rash (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)
skin irritation (Skin and subcutaneous tissue disorders) | 3 (3) | 2 (2)
hematoma evacuation (Surgical and medical procedures) | 0 (0) | 2 (2)
thrombectomy (Surgical and medical procedures) | 0 (0) | 4 (4)
deep vein thrombosis (Vascular disorders) | 0 (0) | 5 (5)
venous thrombosis (Vascular disorders) | 0 (0) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days